CLINICAL TRIAL: NCT05913518
Title: Training Metacognition by Means of Neurofeedback in Subjects With Alcohol Use Disorder Induces Neural Modifications: an Event-related Potentials Study
Brief Title: Neurofeedback Training of Metacognition in Subjects With Alcohol Use Disorder. Disorder Induces Neural Modifications: an Event-related Potentials Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Salvatore Campanella, FNRS Research Director, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Neurofeedback
Record Dates: First submitted 2023-06-01; First posted 2023-06-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active neurofeedback group (Experimental)
  Interventions: Device: Neurofeedback active
- Placebo feedback group (Placebo Comparator)
  Interventions: Device: Neurofeedback placebo
- Control group (No Intervention)

INTERVENTIONS:
Device: Neurofeedback active — Neurofeedback uses real-time displays of brain activity to teach self regulation of brain function. People can learn to control their own brain activity through operant conditioning, where they receive feedback on their brainwaves and learn to modify them to achieve a desired state. Active neurofeedback group aims at enhancing the sensorimotor rhythm (12-15 Hz).
  Arms: Active neurofeedback group
Device: Neurofeedback placebo — Neurofeedback uses real-time displays of brain activity to teach self regulation of brain function. People can learn to control their own brain activity through operant conditioning, where they receive feedback on their brainwaves and learn to modify them to achieve a desired state. Placebo feedback group (PFT) : patients enhance random frequency bands
  Arms: Placebo feedback group

SUMMARY:
Addressing cognitive deficits in alcohol use disorder (AUD) supports recovery. Impaired metacognitive functioning in AUD causes compromised recognition of the interoceptive state leading to the maintenance of alcohol abuse despite negative consequences. By promoting greater self-awareness and self-regulation, neurofeedback training is of high relevance in metacognition remediation to support abstinence.

The main objective of the present study is to validate neurofeedback as a complementary clinical tool to overcome metacognitive deficits that represent a significant factor in the maintenance of harmful consumption behavior and relapse phenomena in AUD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old undergoing a 3- to 4-week detoxification treatment program at the Alcohol Unit of CHU Brugmann hospital (Brussels, BELGIUM), who have been diagnosed with severe AUD (alcohol use disorder) according to the DSM-V-TR.

Exclusion Criteria:

* history of neurological disorders
* other serious medical conditions
* neuroleptic treatment are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Event related potential | Baseline T0
  Error related negativity (ERN) measurement
Event related potential | Immediately after the last neurofeedback training session T1
  Error related negativity (ERN) measurement
Metacognition questionnaire-30 (MCQ-30) | Baseline T0
  Metacognitive assessment by means of a questionnaire. Scores from 6 to 24, with higher scores meaning worse outcomes.
Metacognition questionnaire-30 (MCQ-30) | Immediately after the last neurofeedback training session T1
  Metacognitive assessment by means of a questionnaire. Scores from 6 to 24, with higher scores meaning worse outcomes.

SECONDARY OUTCOMES:
Commission error rate | Baseline T0
  Behavior assessment
Commission error rate | Immediately after the last neurofeedback training session T1
  Behavior assessment
Reaction times | Baseline T0
  Behavior assessment
Abstinence | Immediately after the last neurofeedback training session T1
  Number of days of abstinence
Abstinence | 2 weeks post discharge
  Number of days of abstinence
Abstinence | 1 month post discharge
  Number of days of abstinence
Abstinence | 2 months post discharge
  Number of days of abstinence
Abstinence | 3 months post discharge
  Number of days of abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Campanella, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No